CLINICAL TRIAL: NCT06822114
Title: Substance Balance of [14C]ET-26 in Healthy Chinese Subjects
Brief Title: Substance Balance Trial of Methoxyethyl Etomidate Hydrochloride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ET-26-HCL-CP-001
Record Dates: First submitted 2025-01-25; First posted 2025-02-12 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Methoxyethyl Etomidate Hydrochloride
  Interventions: Drug: Methoxyethyl Etomidate Hydrochloride

INTERVENTIONS:
Drug: Methoxyethyl Etomidate Hydrochloride — The dose is 50 μCi/48 mg，in the fasting state, a single intravenous injection was given slowly

SUMMARY:
This study was a single-center, single-dose, open-label design with 6-8 healthy adult male subjects to evaluate the body material balance of [14C]ET-26. Each subject received a single intravenous injection of [14C]ET-26 at a dose of 50 µCi/48 mg. Blood, urine, and stool samples were collected at specified times during the study. The pharmacokinetic parameters were calculated, and the distribution of total radioactivity in venous whole blood and plasma was analyzed. The excretion rate and pathway were analyzed. The metabolic pathway and elimination pathway of ET-26 in human body were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. healthy Chinese men;
2. The age of signing the informed consent: 18-45 years old;
3. Body mass index of 19-26 kg/m2, body weight of 60 kg±5kg;
4. fully understand the purpose and requirements of the study, and voluntarily sign the informed consent;
5. Able to communicate well with investigators and complete the trial according to the protocol.

Exclusion Criteria:

-

Auxiliary examination:

1. Those with clinically significant abnormalities in comprehensive physical examination, vital signs, laboratory tests, serum cortisol, 12-lead electrocardiogram, chest X-ray, digital anal examination, abdominal ultrasound ;
2. potentially difficult airway ;
3. resting corrected QT interval (QTcF) > 450 ms obtained by 12-lead electrocardiogram;
4. hepatitis B surface antigen or E antigen, hepatitis C virus antibody IgG , or treponema pallidum antibody testing, human immunodeficiency virus antigen/antibody combination testing ;
5. those who are not suitable for arterial blood sampling, such as Allen's test positive;

   Medication history:
6. patients who had taken any prescription drugs, over-the-counter drugs, Chinese herbal medicine, or food supplements from 14 days before screening to the time of drug administration;
7. Use of any drugs that inhibit or induce liver drug enzymes or affect the body's cortisol level between 30 days before screening and before drug administration;

   History of disease and surgery:
8. patients with a history of any clinically serious disease or disease or condition considered by the investigators to be likely to affect the results of the trial, including but not limited to a history of cardiovascular, respiratory, endocrine, nervous, digestive, urinary, or hematologic, immune, psychiatric, or metabolic diseases;
9. patients with a history of adrenal insufficiency, adrenal tumors, or hereditary heme biosynthesis disorders;
10. patients with anesthetic accident history, malignant high fever history or related family history;
11. previous history of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, ventricular tachycardia, atrioventricular block, long QT syndrome or symptoms of long QT syndrome and family history ;
12. had a history or current respiratory disease, including respiratory insufficiency, obstructive lung disease, asthma, or bronchospasm requiring treatment within 3 months before screening; Or acute respiratory infection within one week before screening, with obvious symptoms such as fever, wheezing, nasal congestion and cough;
13. patients who underwent major surgery within 6 months prior to screening or who had incompletely healed surgical incisions, including but not limited to any surgery with a significant risk of bleeding, prolonged general anesthesia, or open biopsy or significant traumatic injury;
14. allergic constitution, such as known allergic history to two or more substances; Or who, as judged by the investigator, may be allergic to the trial drug or its excipients;
15. patients with hemorrhoids or perianal diseases with regular/ongoing hematochezia, gastroesophageal reflux disease, irritable bowel syndrome, inflammatory bowel disease;

    Living habits:
16. habitual constipation or diarrhea;
17. were heavy drinkers or regular drinkers in the 6 months before screening, i.e., drank more than 14 units of alcohol per week (1 unit =360 mL of beer, 45 mL of 40% spirits, or 150 mL of wine), had an alcohol breath test ≥20 mg/dl at screening, or were unable to abstain from alcohol during the trial;
18. smoked more than 5 cigarettes per day or were habitual users of nicotine-containing products in the 3 months before screening, or were unable to quit during the trial;
19. abusing drugs or using soft drugs 3 months before screening or hard drugs 1 year before screening; Or positive urine drug test during screening period;
20. habitual drinkers of grapefruit juice or excessive tea, coffee and/or caffeinated beverages who were unable to abstain during the trial;
21. with strenuous exercise and other factors affecting drug absorption, distribution, metabolism and excretion;

    Others:
22. workers who are exposed to radioactive conditions for a long time, or have had significant radiation exposure within 1 year before screening, or participated in radiopharyngology labeling tests;
23. patients with a history of syncope, or difficulty in blood collection, or can not tolerate venipuncture blood collection;
24. those who had taken any investigational drug or used any investigational device within 3 months before screening;
25. vaccinated within 1 month before screening or planned to be vaccinated during the trial period;
26. had plans to give birth or donate sperm within 1 year after signing the informed consent form, or did not agree to take strict contraceptive measures for the subjects and their spouses within 1 year after completing the study ;
27. if they had lost blood or donated ≥400 mL within 3 months before screening, received a transfusion or blood component within 1 month, or were planning to donate blood during the trial;
28. those who have special requirements for diet or cannot abide by the uniform diet; Or they refused to discontinue any beverage containing xanthine derivatives such as caffeine for 48 hours before drug administration until the end of the study; The subjects refused to stop eating animal offal, seafood, soy products and other foods with high purine content.
29. had any other factors considered by the investigator to preclude participation in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic parameters | Up to 168 hours after drug administration.
  Cmax

SECONDARY OUTCOMES:
MOAA/S score | Up to 20 minutes after drug administration.
  modified observer's assessment of alert（MOAA/S） score: The lowest score was 0, indicating full anesthetic sedation, and the highest score was 5, indicating full consciousness.

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, Doctor, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China